CLINICAL TRIAL: NCT00904579
Title: Cancer Risk in Solid Organ Transplant Recipients and End-Stage Renal Disease: The Transplant Cancer Match Study
Brief Title: Cancer Risk in Organ Transplant Recipients and End-Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906194; 06-C-N194; NCT01445574 (obsolete NCT alias)
Record Dates: First submitted 2009-05-16; First posted 2009-05-19 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Immunocompromised Host; Organ Transplantation; Cancer
Keywords: Organ Transplants; Immunosuppression; Cancer; End Stage Renal Disease; ESRD; Cancer Risk
MeSH Terms: conditions — Neoplasms; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Cancer patients who have had organ transplants identified through the transplant and cancer registries.

SUMMARY:
Background:

* Solid organ transplantation provides life-saving treatment for end-stage organ disease but is associated with an increased cancer risk because of the need for long-term immunosuppression
* End-stage renal disease (ESRD), the most common type of end-stage organ disease leading to transplant, is itself linked to increased risk for some cancers
* The role of immunosuppression and other factors causing cancer in this setting are not fully understood.

Objectives:

* To characterize cancer risk in transplant recipients and identify risk factors.
* To characterize risk for transmission of cancer from organ donors to recipients.
* To describe cancer risk in ESRD.

Eligibility: Patients are not required for this study. Data are gathered from existing databases of ESRD patients, organ transplant patients and cancer registries.

Design:

* Databases of 1) U.S. transplant recipients, donors and wait list candidates and 2) U.S. ESRD patients will be linked to multiple U.S. cancer registries to identify cancers in transplant recipients and ESRD patients.
* The spectrum of cancer risk in transplant recipients and ESRD patients will be evaluated in detail.
* The cancer risk in transplant recipients will be examined in relation to whether the donors had cancer.
* The proposed cancer risk factors (e.g., underlying medical condition, infection with cancer-causing viruses, immunosuppressive medications) documented in transplant and ESRD files will be studied for association with increased risk of particular types of cancer.

DETAILED DESCRIPTION:
Solid organ transplantation provides life-saving treatment for end-stage organ disease but is associated with substantially elevated cancer risk, largely due to the need to maintain long-term immunosuppression. Despite previous research, important research questions remain concerning the role of immunosuppression and other factors in causing cancer in the setting. Staff at two federal agencies, the National Cancer Institute (NCI) and the Health Resources and Services Administration (HRSA), will link a database containing information on U.S. transplant recipients, wait list candidates, and donors to multiple U.S. cancer registries. These data will be used to conduct research concerning the spectrum of cancer risk in transplant recipients. The data will also be used by HRSA in its public health role overseeing the U.S. solid organ transplant network to maintain and improve safety of organ transplantation.

ELIGIBILITY:
* This study will include as subjects all individuals included in the transplant data set. All U.S. solid organ transplant recipients, candidates for transplant, and living related donors.

In addition, the study will include all individuals in the U.S. ESRD data set.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients who have had organ transplants identified through the transplant and cancer registries.@@@
Sampling Method: Non-Probability Sample
Enrollment: 19929901 (Estimated)
Dates: Start 2006-07-01 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Cancer | End of study
  Cancer patients who have had organ transplants identified through the transplant and cancer registries.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Engels, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- United States (9):
  - California Cancer Registry, Sacramento, California
  - Colorado Cancer Registry, Denver, Colorado
  - Connecticut Cancer Registry, Hartford, Connecticut
  - Georgia Cancer Registry, Atlanta, Georgia
  - Iowa Cancer Registry, Iowa City, Iowa
  - National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland
  - New Jersey Cancer Registry, New Brunswick, New Jersey
  - New York Cancer Registry, Albany, New York
  - Seattle Cancer Registry, Seattle, Washington